CLINICAL TRIAL: NCT04954144
Title: The Effect of Fine Motor Grip Studies in Virtual Reality Environment on Performance-Based Hand Skills in Children With Cerebral Palsy
Brief Title: Role of Virtual Reality in Hand Rehabilitation for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ayşe Neriman NARİN, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-ANN-01
Record Dates: First submitted 2021-04-26; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Physical Disability; Cerebral Palsy
Keywords: cerebral palsy; virtual rehabilitation; hand rehabilitation; leap motion
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leap Motion Sensor (Experimental): The Leap Motion Sensor is an optical hand tracking module that captures the movements of hands with unparalleled accuracy.
  Interventions: Device: Leap Motion Sensor; Other: Neurodevelopmental Treatment Approach
- Neurodevelopmental Treatment Approach (Experimental): Neurodevelopment treatment approach is used to influence the quality of the motor response and is carefully matched to the patient's abilities to use sensory information and adapt movements.
  Interventions: Other: Neurodevelopmental Treatment Approach

INTERVENTIONS:
Device: Leap Motion Sensor — As a virtual reality treatment method, leap motion sensor was integrated with laptop computer and participants played object capture, firefly, bee-batting games to improve performance based hand skills.
  Arms: Leap Motion Sensor
Other: Neurodevelopmental Treatment Approach — It is a method that tries to control sensorimotor components of muscle tone, reflexes, abnormal movement patterns, postural control, sensory-perception and memory problems with special techniques.

SUMMARY:
Cerebral Palsy (CP) is a neurodevelopmental dysfunction which is permanent, non-progressive, and caused by brain insult or injury.Although the basic finding of CP is having motor function problems, visual, auditory, cognitive and behavioural problems are also seen in CP.Having these problems interfere the functional independence of children with CP, so their daily life of activities is limited.One of the way of increasing the functional independence of these children is providing them hand rehabilitation.In the event of having hand rehabilitation, children would achieve more daily living skills.Although having hand rehabilitation is crucial for these children, they would lose their motivation on this by the time because rehabilitation is a long process,For that reason, new therapy techniques are tried by therapists to motivate these children during their rehabilitation seances.Virtual reality rehabilitation is one of these new techniques used for designing enjoyable and effective seances.Especially leap motion sensors are preferred to create virtual environment, because they are cheap, portable, touchless and easy to use.These sensors can detect hand movements and recognize hand gestures by using infrared.Our study was aimed to investigate the effect of fine motor grip studies in virtual reality environment on performance based hand skills in children with CP.Thirty two children with CP (6-18) were included in this study.Children were randomly assigned into two equal-sized groups: control and study groups.Participants in both groups received a neurodevelopmental therapy program.The study group additionally received virtual reality rehabilitation programme. In control group, neurodevelopmental treatment was provided 45 mins,2 d/week for 2 successive months.In study group, neurodevelopmental treatment was provided 30 mins and virtual rehabilitation programme was provided 15 mins, 2 d/week for 2 successive months. To evaluate the performance based hand skills; Box and Block Test, Nine Hole Peg Test and Pink Tower (Montessori) Test were used.

DETAILED DESCRIPTION:
Cerebral palsy (CP) can be defined as a permanent, non-progressive, motor function, posture and developmental disorder that causes movement limitation due to a lesion that can occur in the brain due to prenatal, perinatal and postnatal reasons.Although the etiology of the disease cannot be determined precisely, the reasons causing SP; It is stated that it occurs in prenatal, perinatal and postnatal periods. Sometimes, more than one factor can be found together.Another common problem in individuals with CP is seen in upper extremity functions, and limiting upper extremity functions also affects the independence of daily living activities. The condition of the hand in the early period of rehabilitation has an important place for upper extremity functions in the future.In this respect, it is very important to include a program to develop manual skills in the rehabilitation process in order to make children with CP more independent in daily life activities.Neurodevelopmental Treatment Approach, widely used in the treatment of children with Cerebral Palsy; It is a method that tries to control sensorimotor components of muscle tone, reflexes, abnormal movement patterns, postural control, sensory-perception and memory problems with special techniques.Virtual reality is a three-dimensional simulation that makes you feel to be in any "place" and provides this by giving various inputs to our sensory organs. According to motor control and motor learning theory, it is important to carry out repetitive, target-oriented studies that increase motivation in the rehabilitation of children with Cerebral Palsy and it is important to include games and entertainment in the treatment program. To achieve this, making virtual reality a component of rehabilitation can cause the treatment process to be more functional and effective.Research has shown that computer games designed for a specific purpose can increase the motivation of children to increase the use of the affected extremities and positively improve the strength and functionality of the affected muscles.Leap Motion Sensors have been developed to detect hand movements. It can detect the movement of the hand by emitting infrared rays in a restricted area. Physiotherapists have stated that virtual reality rehabilitation applied with Leap Motion Sensors can be an effective method that increases motivation in the treatment process in children with special needs.Our study was aimed to investigate the effect of fine motor grip studies in virtual reality environment on performance based hand skills in children with CP.After the approval of the ethics committee, children with cerebral palsy were included in the study.Parental approval was obtained.Reports from Health Council was examined to check diagnosis of children.The study was performed in three centers: University of Abant Izzet Baysal, Silivri Rehabilitation Center and Reyhan Rehabilitation Center.Thirty two children with CP (6-18) were included in this study.Exclusion criteria were; epilepsy history, cognitive problems, visual impairment, having problem on holding and releasing the objects.Children were randomly assigned into two equal-sized groups: control and study groups.Participants in both groups received a neurodevelopmental therapy program.The study group additionally received virtual reality rehabilitation programme.As a normal developmental treatment method, functional skills exercises, inhibition of abnormal movement patterns, sensory-motor integration in purposeful movements, stretching and strengthening exercises, and daily life activities were trained.As a virtual reality treatment method, object catching, firefly, bee-batting games were used, which improved performance-dependent dexterity by integrating leap motion sensors into the laptop.In control group, neurodevelopmental treatment was provided 45 mins,2 days/week for 2 successive months.In study group, neurodevelopmental treatment was provided 30 mins and virtual rehabilitation programme was provided 15 mins, 2 days/week for 2 successive months.In virtual reality treatment, each game was studied for 5 minutes and 3 games for a total of 15 minutes.Before and after the study, tests that measure performance-related dexterity were applied and the previous and next results of the groups were compared.SPSS statistics program was used for statistical evaluation of data belonging to participants.In statistical evaluations, p <0.05 was considered as significant.In the data analysis of the study, in order to select the appropriate statistical analysis, whether the distribution of the data is suitable for normal distribution was determined by the "one-sample Kolmogorov-Smirnov" test."Independent T Test" was used to compare age, height, body weight, the measures pre-treatment and post-treatment, .Gender and affected sides were compared by using "Chi-Square Test".

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Functional Level should be I or II.

Exclusion Criteria:

* Epilepsy
* Visual Impairment
* Cognitive Problem
* Inability to hold and release the objects

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
ABILHANDS-kids Scoring Before Study | Day 1
  Measure of manual ability for children with upper limb impairments before study.
ABILHANDS-kids Scoring After Study | Day 56
  Measure of manual ability for children with upper limb impairments after study.
Manual Ability Classification System | Day 1
  It describes how children with cerebral palsy use their hands to handle objects in daily activities.
Gross Motor Function Classification | Day 1
  It description of a child's current motor function
Box and Block Test Before Study | Day 1
  It measures unilateral gross manual dexterity before study.
Box and Block Test After Study | Day 56
  It measures unilateral gross manual dexterity after study.
9 Hole Peg Test Before Study | Day 1
  It is a standardized, quantitative assessment used to measure finger dexterity before study.
9 Hole Peg Test After Study | Day 56
  It is a standardized, quantitative assessment used to measure finger dexterity after study.
Pink Tower Montessori Test Before Study | Day 1
  It measures performance based hand skill before study.
Pink Tower Montessori Test After Study | Day 56
  It measures performance based hand skill after study.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Neriman Narin, Asst.Prof, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Silivri Rehabilitation Center, Istanbul, Silivri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No